CLINICAL TRIAL: NCT05051332
Title: A Multi-Center, Active-Controlled, Open-Label, Phase III Trial to Compare the Efficacy and Safety for Treatment of Autologous Chondrocytes Implantation With CartiLife Versus Microfracture for Patients With Knee Chondral Defects
Brief Title: Phase 3 Clinical Trial of CartiLife® in Korea
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Biosolution Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BS-CTL-III
Record Dates: First submitted 2021-08-04; First posted 2021-09-21 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2021-09

CONDITIONS: Articular Cartilage Defect; Articular Cartilage Degeneration

STUDY DESIGN:
Intervention Model Description: Investigational Group : CartiLife® Procedure: Extracellular matrix-associated autologous chondrocytes comprise CartiLife®, composed as pellets (1.1 to 1.8 mm in diameter) in suspension. One pre-filled syringe is implanted per 1 cm^3 of defect volume, and fibrin adhesive is applied to fix pellets in place through minimal arthrotomy.
  Active comparator: Microfracture Surgery Procedure : Microfracture surgery, performed by arthroscopy after the joint is cleaned of calcified cartilage, will be conducted using an awl or drill to create tiny fractures in the subchondral bone plate.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CartiLife® (Experimental): Extracellular matrix-associated autologous chondrocytes comprise CartiLife®, composed as pellets (1.1 to 1.8 mm in diameter) in suspension. One pre-filled syringe is implanted per 1 cm^3 of defect volume, and fibrin adhesive is applied to fix pellets in place through minimal arthrotomy.
  Interventions: Drug: Autologous Chondrocyte Implantation (CartiLife®)
- Microfracture Surgery (Active Comparator): Microfracture surgery, performed by arthroscopy after the joint is cleaned of calcified cartilage, will be conducted using an awl or drill to create tiny fractures in the subchondral bone plate.
  Interventions: Procedure: Microfracture Surgery

INTERVENTIONS:
Drug: Autologous Chondrocyte Implantation (CartiLife®) — CartiLife consists of small beads (1 mm in diameter) in suspension, developed from pellet culture of autologous costal chondrocytes after multiplication. The beads are implanted in an injective manner with fibrin glue through minimal arthrotomy. The dose depends on the size (volume) of the defect, recommended dose is 480 pellets/cm^3 defect
  Other Names: CartiLife
  Arms: CartiLife®
Procedure: Microfracture Surgery — Microfracture surgery, performed by arthroscopy after the joint is cleaned of calcified cartilage, will be conducted using an awl or drill to create tiny fractures in the subchondral bone plate
  Arms: Microfracture Surgery

SUMMARY:
To evaluate the safety and efficacy of pellet-type extracellular matrix-associated autologous chondrocytes (CartiLife®) obtained by cultivating costal chondrocytes of the subject implanted into articular cartilage defects of the knee resulting from trauma or degeneration.

DETAILED DESCRIPTION:
This open-label, phase 3 study is being conducted to evaluate the safety and efficacy of pellet-type extracellular matrix-associated autologous chondrocytes (CartiLife®) compared with microfracture surgery in adults with articular cartilage defects due to trauma or degeneration of the knee. It is hypothesized that CartiLife® treatment will demonstrate structural regeneration and improvement in function and pain at Week 48 compared to baseline.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, an individual must meet all of the following:

1. Patients over the age of 18.
2. Defect size: 2 to 10 cm^2 on the unilateral knee cartilage (up to 4 ㎤ in volume).
3. Defect: isolated ICRS (International Cartilage Repair Society) grade III or IV single defect chondral lesion on articular cartilage with comparatively healthy cartilage present near the lesion site (ICRS Grade 1 ~ 2).
4. Patients with a KOOS total score below 55.
5. Patients able to walk without aid.
6. Patients who agree to abide by rehabilitation protocols and follow-up programs, including residential exercise routines.
7. Patients who provide written consent to the application of the clinical trial.

Exclusion Criteria:

Individuals who meet any of the following will be excluded from participation in this study:

1. Patients with inflammatory articular diseases such as rheumatoid arthritis or gouty arthritis.
2. Patients scoring 3 or above on the Kellgren-Lawrence Grading Scale.
3. Patients with inflammatory articular diseases related to autoimmune diseases.
4. Patients hypersensitive to bovine derived proteins or any of the components in this product.
5. Patients hypersensitive to Gentamycin.
6. Patients with Haemophilia or markedly reduced immune function.
7. Patients with arterial bleeding and severe venous bleeding.
8. Patients with other diseases including tumors except for cartilaginous defects of joints.
9. Patients with a history of radiation treatment and chemotherapy within the past two years.
10. Patients who are pregnant, or nursing a baby.
11. Patients who participate in concurrent clinical trials or previous clinical trials within 30 days of administration.
12. Other cases where the investigator deems the patient ineligible for participation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2020-03-19 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
MOCART (Magnetic Resonance Observation of Cartilage Repair Tissue) | At Week 48, post-operation
  MOCART is a validated tool that provides reliable, reproducible, and accurate assessment of cartilage repair tissue (Marlovits et al, 2006 that; Trattnig et al, 2011).
KOOS Total Score | From Week 0 to Week 48, post-operation
  The KOOS is a reliable and valid patient-reported outcome measurement tool that evaluates both short-term and long-term consequences of knee injury. The 5 separately scored subscales of Pain, other Symptoms, Function in daily living (ADL), Function in Sport and Recreation (Sport/Rec), and knee-related QOL may enrich clinical and research data interpretation (Roos and Lohmander, 2003; Collins et al, 2011).
  In the 'Knee injury and Osteoarthritis Outcome Score', scores range from 0 to 100 with a score of 0 indicating the worst possible knee symptoms and 100 indicating no knee symptoms.

SECONDARY OUTCOMES:
MOCART Score | At Week 24 and Week 96, post-operation
  MOCART is a validated tool that provides reliable, reproducible, and accurate assessment of cartilage repair tissue (Marlovits et al, 2006 that; Trattnig et al, 2011).
  In the 'Magnetic Resonance Observation of Cartilage Repair Tissue (MOCART) Score', the total score ranges from 0 to 100, with a score of 0 indicating the worst possible knee symptoms and 100 indicating no knee symptoms.
Lysholm Score | At Week 0 to Week 8, 24, 48 and 96, post-operation
  The Lysholm scale is a broadly applicable, validated tool for measuring changes following nonsurgical and surgical intervention, as well as deterioration over time in patients with various knee pathologies (Collins et al, 2011).
  In the 'Lysholm score', the total score ranges from 0 to 100, with a score of 0 indicating the worst possible knee symptoms and 100 indicating no knee symptoms.
IKDC Score | At Week 0 to Week 8, 24, 48 and 96, post-operation
  The IKDC Knee form covers domains likely to be important to patients and has adequate consistency and broad applicability across mixed groups of patients (Collins et al, 2011).
  In the 'International Knee Documentation Committee Subjective Knee Form', the total score ranges from 0 to 100, with a score of 0 indicating the worst knee symptoms(lowest level of function or highest level of symptoms) and 100 indicating no knee symptoms(highest level of function and lowest level of symptoms).
KOOS Score (Pain, Other symptoms, Function in daily living, Function in sport and recreation, and knee-related QOL subscales) | At Week 0 to Week 8, 24, 48 and 96, post-operation
  The KOOS is a reliable and valid patient-reported outcome measurement tool that evaluates both short-term and long- term consequences of knee injury. The 5 separately scored subscales of Pain, other Symptoms, Function in daily living (ADL), Function in Sport and Recreation (Sport/Rec), and knee-related QOL may enrich clinical and research data interpretation (Roos and Lohmander, 2003; Collins et al, 2011).
  KOOS Score (Pain, Other symptoms, Function in daily living, Function in sport and recreation, and knee-related QOL subscales) are measured between 0, 1, 2, 3 and 4. The KOOS subscales are scored separately: Pain (9 items); Symptoms (7 items); Function in daily living (17 items); Function in sport and recreation (5 items); knee-related QOL (4 items). Each scale is scored between 0 to 4. The total score ranges from 0 to 100, with a score of 0 indicating the worst possible knee symptoms and 100 indicating no knee symptoms.
VAS (100mm Pain Visual Analogue Scale) | At Week 0 to Week 8, 24, 48 and 96, post-operation
  The VAS is a validated, ubiquitous tool for patient-reported measurement of pain at a given point in time (Kersten et al, 2014).
  Visual Analogue Scale (VAS) is a measurement instrument that measures a specified characteristic which is deemed difficult to quantify across a continuous line of value to determine its representative value. The VAS scale ranges from 0 to 100 mm, with 0 indicating absence of pain and 100 indicating the worst pain experienced.
Tegner Activity Scale | At Week 0 to Week 8, 24, 48 and 96, post-operation
  The Tegner activity score is a frequently used patient-administered activity rating system for patients with various knee activity functions. The instrument scores a person's activity level between 0 and 10 where 0 is 'on sick leave/disability' and 10 is 'participation in competitive sports such as soccer at a national or international elite level' (Karen Hambly, 2011). A level of 0 indicates that the patient is unable to participate in activities barring 'Sick leave or disability pension because of knee problems', and a level of 10 indicates that the patient is capable of participating in activities which at its most intense include 'Competitive sports - soccer, football, rugby at a national elite level'.
Pain medication history | At Week 0 to Week 8, 24, 48 and 96, post-operation
  Pain medication history is an indicator of patient pain. Pain medication history is an indicator of patient pain. The frequency of analgesic ingestion is measured for the specified duration over the course of the clinical trial, and changes in analgesic ingestion in terms of frequency are assessed to analyze the efficacy of the clinical trial product.
Treatment related adverse events | At Week 0 (pre-operation), and up to 24 Months (post-operation)
  Number of subjects with treatment related adverse events as assessed by analysis of adverse events including symptoms, abnormal findings on physical examination, vital signs, ECG, and standard laboratory examination results. The total number of patients who exhibit symptoms identified as an adverse event will be cumulatively combined to obtain a whole digit number representing the number of patients who have suffered an adverse event throughout the course of the clinical trial.

CONTACTS AND LOCATIONS:
Overall Officials: Jungsun Lee, Ph.D, Study Director — Biosolution Co., Ltd.; Kyoung Ho Yoon, MD, Principal Investigator — Kyung Hee University Hospital; Jae Doo Yoo, MD, Principal Investigator — Ewha Womans University Mokdong Hospital; Sang Hak Lee, MD, Principal Investigator — Kyung Hee University Hospital at Gangdong; Sung-Hwan Kim, MD, Principal Investigator — Gangnam Severance Hospital; Ji Hoon Bae, MD, Principal Investigator — Korea University Guro Hospital; Hyuk-Soo Han, MD, Principal Investigator — Seoul National University Hospital; Joon Ho Wang, MD, Principal Investigator — Samsung Medical Center; Min Jung, MD, Principal Investigator — Severance Hospital; Yong In, MD, Principal Investigator — The Catholic UNIV. of Korea Seoul St. Mary's Hospital; Chong Bum Chang, MD, Principal Investigator — Seoul National University Bundang Hospital (1); Yong Seuk Lee, MD, Principal Investigator — Seoul National University Bundang Hospital (2); Seok Jung Kim, MD, Principal Investigator — The Catholic UNIV. of Korea Uijeongbu St. Mary's Hospital; Jong Geun Seon, MD, Principal Investigator — Chonnam National University Hospital; Dong Hwi Kim, MD, Principal Investigator — Chosun University Hospital; Young-Mo Kim, MD, Principal Investigator — Chungnam National University Hospital; Seung Joon Rhee, MD, Principal Investigator — Pusan National University Hospital; Sang Won Moon, MD, Principal Investigator — Haeundae Paik Hospital, Inje University; Young Choi, MD, Principal Investigator — Kosin University Gospel Hospital
Locations (18):
- South Korea (18):
  - Inje University Haeundae Paik Hospital, Busan
  - Kosin University Gospel Hospital, Busan
  - Chungnam National University Hospital, Daejeon
  - Chonnam National University Hwasun Hospital, Gwangju
  - Chosun University Hospital, Gwangju
  - Pusan National University Hospital, Pusan
  - Seoul National University Bundang Hospital (1), Seongnam-si
  - Seoul National University Bundang Hospital (2), Seongnam-si
  - Kyung Hee University Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Kyung Hee University Hospital at Gangdong, Seoul
  - Gangnam Severance Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Ewha Womans University Mokdong Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - The Catholic UNIV. of Korea Seoul St. Mary's Hospital, Seoul
  - The Catholic UNIV. of Korea Uijeongbu St. Mary's Hospital, Uijeongbu-si

IPD SHARING:
Plan to Share IPD: No
There are no future plans to share the IPD at this time.

REFERENCES:
- [Background] Yoon KH, Park JY, Lee JY, Lee E, Lee J, Kim SG. Costal Chondrocyte-Derived Pellet-Type Autologous Chondrocyte Implantation for Treatment of Articular Cartilage Defect. Am J Sports Med. 2020 Apr;48(5):1236-1245. doi: 10.1177/0363546520905565. Epub 2020 Mar 3. PMID 32125878
- [Background] Yoon KH, Yoo JD, Choi CH, Lee J, Lee JY, Kim SG, Park JY. Costal Chondrocyte-Derived Pellet-Type Autologous Chondrocyte Implantation versus Microfracture for Repair of Articular Cartilage Defects: A Prospective Randomized Trial. Cartilage. 2021 Dec;13(1_suppl):1092S-1104S. doi: 10.1177/1947603520921448. Epub 2020 Jun 1. PMID 32476445
- Available data/document: Clinical Study Report: NCT03545269 — https://clinicaltrials.gov/ — Study to Assess the Efficacy and Safety of Treatment of Articular Cartilage Lesions With CartiLife®
- Available data/document: Clinical Study Report: NCT03517046 — https://clinicaltrials.gov/ — Study to Assess the Safety of Treatment of Articular Cartilage Lesions With CartiLife®